CLINICAL TRIAL: NCT05917613
Title: Complex-Posttraumatic Stress Disorder - Cultural Adaptation of a Therapeutic Manual and Development of a Culture-specific Diagnostic Module for Refugee Populations in Switzerland (Pilot Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Heim (Other)
Responsible Party: Sponsor-Investigator, Eva Heim, Associate professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00464
Record Dates: First submitted 2023-05-13; First posted 2023-06-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Complex Post-Traumatic Stress Disorder

STUDY DESIGN:
Intervention Model Description: Pilot
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Psychotherapy
  Interventions: Behavioral: Enhanced Skills Training in Affective and Interpersonal Regulation combined with Modified Prolonged Exposure (ESTAIR/MPE)

INTERVENTIONS:
Behavioral: Enhanced Skills Training in Affective and Interpersonal Regulation combined with Modified Prolonged Exposure (ESTAIR/MPE) — Psychotherapeutic manual for the treatment of Complex Post-Traumatic Stress Disorder (CPTSD)

SUMMARY:
In January 2022, the World Health Organization (WHO) launched the 11th edition of the International Classification of Diseases (ICD-11). This diagnostic manual includes the new diagnosis of complex post-traumatic stress disorder (CPTSD). This new diagnostic category describes difficulties that may arise as a result of multiple, prolonged or repeated trauma, from which it is difficult or impossible to escape, such as torture, domestic violence or childhood sexual abuse. People affected by CPTSD often have difficulty regulating their emotions and maintaining relationships with others, and they often show a negative self-concept.

Evidence from the field of cultural clinical psychology indicates cultural variation in the CPTSD symptoms across different cultural groups. In addition, psychopathology is shaped by structural factors such as inequality and/or discrimination.

This research project aims to highlight such cultural and structural aspects related to PTSD and CPTSD among refugee populations in Switzerland. A diagnostic interview and a therapeutic manual will be culturally adapted and pilot tested with a small sample (n = 24).

ELIGIBILITY:
Inclusion Criteria:

* Refugees and asylum seekers from the greater Middle Eastern and Northern Africa (MENA) region, regardless of their residence permit. The four languages that will be used for the planned project are: Farsi/Dari, Arabic, Turkish, and Kurdish (Kurmanji).
* "High risk" (i.e., minimally 8 points) on the questionnaire Process of Recognition and Orientation of Torture Victims in European Countries to facilitate Care and Treatment (PROTECT);
* age 18 or older;
* informed consent signed

Exclusion Criteria:

* imminent risk of suicide;
* acute psychosis;
* severe alcohol and/or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility ESTAIR manual | 7 months
  Feasibility of the ESTAIR manual will be evaluated via the percentage of users who who adhere to the therapy until the end (out of those who start the therapy). As general rule, 80-90% adherence is considered as excellent, 70-80% as satisfactory, and 60-70% as acceptable.
Feasibility International Trauma Interview (ITI) | 1 month
  Feasibility will be examined based on the percentage of participants who complete the ITI. As general rule, 80-90% participation and adherence is considered as excellent, 70-80% as satisfactory, and 60-70% as acceptable.
Feasibility research procedures | 7 months
  Feasibility will be evaluated based on the percentage of participants who give their informed consent (out of those invited) and based on the percentage of participants who adhere to the study until the end (out of those who sign the informed consent). As general rule, 80-90% participation and adherence is considered as excellent, 70-80% as satisfactory, and 60-70% as acceptable.
Acceptability International Trauma Interview (ITI) | 1 month
  Acceptability of the ITI will be assessed through qualitative interviews after the diagnostic interview. Content analysis will be used to extract the most important information related to acceptability.
Acceptability ESTAIR/MPE | 7 months
  Acceptability will be assessed through the qualitative interviews after each of the four modules. Content analysis will be used to extract the most important information related to acceptability.
Acceptability research procedures | 7 months
  Acceptability of the research procedures will be assessed through qualitative interviews at the end of the study. Content analysis will be used to extract the most important information related to acceptability.

SECONDARY OUTCOMES:
Complex post-traumatic stress disorder | 7 months
  International Trauma Interview. This interview evaluates 12 symptoms (6 for post-traumatic stress disorder and another 6 for disturbances in self-organisation). A diagnosis of complex post-traumatic stress disorder requires that the post-traumatic stress disorder criteria are satisfied (with a diminished startle response if hypervigilance or exaggerated startle are not present), and the endorsement of one of two symptoms from each of the three "disturbances in self-organisation" symptom clusters, plus endorsement of functional impairment associated with these symptoms. Endorsement of a symptom requires that it is trauma related, has been present for at least a year and scores > 2.
Depression | 7 months
  Patient Health Questionnaire (PHQ-9). The PHQ-9 score may range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores mean higher levels of depression.
Anxiety | 7 months
  General Anxiety Disorder Questionnaire (GAD-7). The GAD-7 score may range from 0 to 21, since each of the 7 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores mean higher levels of anxiety.
Somatic Symptoms | 7 months
  Somatic Symptoms Scale (SSS-8). The SSS-8 score may range from 0 to 32, since each of the 8 items can be scored from 0 (not at all) to 4 (severely). Higher scores mean higher levels of anxiety.
Wellbeing | 7 Months
  WHO-5 questionnaire. Scores range from 0-25, with higher scores reflecting higher levels of well-being

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Ambulatorium für Folter- und Kriegsopfer, Wabern, Canton of Bern
  - Appartenances, Lausanne